CLINICAL TRIAL: NCT05558787
Title: Aromatic L-amino Acid Decarboxylase Activity, Tyrosine Decarboxylase Activity and Gut Microbiome in Patients With Advanced Parkinson's Disease
Brief Title: AADC/TDC in Advanced Parkinson's Disease
Acronym: AADCTDC
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: University of Groningen (Other); Predica Diagnostics (Unknown); ParkinsonNL (Unknown); Maag Lever Darm Stichting (Other); Stichting Woelse Waard (Unknown); Stichting Alkemade-Keuls (Unknown)
Responsible Party: Sponsor
Other Study IDs: 113707
Record Dates: First submitted 2022-09-09; First posted 2022-09-28 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Feces, serum, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rationale: Many persons with Parkinson's disease (PD) develop a progressive resistance to levodopa, which is the pharmacological mainstay of PD treatment. Recently, two enzymatic pathways have been identified that could be (partially) responsible for this: 1) breakdown of levodopa by bacterial tyrosine decarboxylase (TDC), an enzyme which normally decarboxylates dietary tyrosine but which is also able to decarboxylate levodopa. Accumulation of bacterial TDC in the small intestine, such as in the context of small-intestinal bacterial overgrowth (SIBO) - for which persons with PD are at increased risk - has the potential to prematurely metabolize levodopa, hence limiting its bioavailability and effect. 2) paradoxical induction of activity of the enzyme aromatic L-amino acid decarboxylase (AADC) in chronic users of levodopa combined with a peripheral decarboxylase inhibitor, also leading to a premature breakdown of levodopa and limitation of its bioavailability and effect.

Primary objective: in a cross-sectional sample of advanced (≥5 years) Parkinson's disease determining the prevalence of increased bacterial TDC activity in feces, and the prevalence of increased AADC activity in serum.

Secondary objective: correlating these biomarkers to clinical parameters, correlating composition of the microbiome to TDC activity, to the presence of levodopa resistance, and to factors related to socio-economic status.

Study design: using feces, serum and urine samples and clinical data from n=50 participants, the relevant enzymes' activity will be measured and the composition of the gut microbiome will be determined. These will be correlated to the clinical and demographic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Participant has Parkinson's disease of at least 5 years duration, defined as time since diagnosis made by a neurologist;
* Participant is an adult, at least 25 years of age;
* Participant can read and understand Dutch;
* Participant has completed the Ethics Committee-approved Informed Consent;
* Participant is willing, competent, and able to comply with all aspects of the protocol, including not taking their PD medication during a 12-hour period, and biospecimen collection.

Exclusion Criteria:

* Co-morbidities that would hamper interpretation of parkinsonian disability, such as coincident musculoskeletal abnormalities, as judged by the investigators;
* Significant doubt over the correctness of the diagnosis PD, as judged by the investigators;
* Not able to stand or walk without the assistance of another person (walking aids are not an exclusion criterion);
* Never having used levodopa;
* No current use of levodopa due to lack of effect, despite never having used at least 600mg/day during at least 1 month;
* Documented allergic reaction or severe side effect to levodopa or benserazide;
* History of narrow-angle glaucoma (unless specific permission by the treating ophthalmologist for use of levodopa/benserazide);
* History of malignant melanoma (unless specific permission by the treating dermatologist for use of levodopa/benserazide);
* History of psychiatric disease with a psychotic component (unless specific permission by the treating psychiatrist for use of levodopa/benserazide);
* Known current uncompensated cardiovascular, endocrine, renal, hepatic, hematologic, or pulmonary disease (unless specific permission by the treating physician for use of levodopa/benserazide);
* Documented severe and debilitating dyskinesias on levodopa, to such an extent that levodopa treatment was terminated;
* Current pregnancy or breastfeeding;
* Co-morbidity with primary gastrointestinal pathology associated with altered gut microbiota and/or altered absorption (such as inflammatory bowel disease, celiac disease, colorectal carcinoma);
* Antibiotic use at any time during the 12 months leading up to the clinic visit;
* Current or recent (less than 1 month before clinic visit) use of (non-parkinson) drugs known or suspected to influence AADC activity, including amphetamine, dexamethasone, dopamine receptor antagonists, monoamine oxidase (MAO) inhibitors (including MAO-B inhibitors which are infrequently used as antiparkinsonian drugs), prostaglandin E2, and vigabatrin.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 adult patients with Parkinson's disease (diagnosed by a neurologist), with a disease duration of at least 5 years (since diagnosis).
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2023-06-28 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2024-08-14 (Actual)

PRIMARY OUTCOMES:
Prevalence of increased TDC activity in feces | through study completion, an average of 2 weeks
Prevalence of increased AADC activity in serum | through study completion, an average of 2 weeks

SECONDARY OUTCOMES:
Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part III | through study completion, an average of 2 weeks
  Baseline score and score after levodopa administration
Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part IV | through study completion, an average of 2 weeks
  Baseline score and score after levodopa administration
Timed up-and-go test | through study completion, an average of 2 weeks
  TUG. Baseline score and score after levodopa administration
Purdue Pegboard Test | through study completion, an average of 2 weeks
  Baseline score and score after levodopa administration
Composite Clinical Motor Score | through study completion, an average of 2 weeks
  This is a composite of MDS-UPDRS-III, TUG and pegboard test scores. Baseline score and score after levodopa administration.
modified Hoehn & Yahr score | through study completion, an average of 2 weeks
  Ordinal scale of Parkinson's disease severity. Baseline score and score after levodopa administration.
9-item Wearing-Off Questionaire (WOQ-9) | through study completion, an average of 2 weeks
  Questionnaire on wearing-off symptoms
SIBO questionnaire | through study completion, an average of 2 weeks
  15-item scale on gastrointestinal symptoms associated with small-intestinal bacterial overgrowth (SIBO)
Schwab and England Activities of Daily Living Scale | through study completion, an average of 2 weeks
  Single-question scale on the ability to perform activities of daily living
Medication questionnaire | through study completion, an average of 2 weeks
  9-item questionnaire on (current and past) medication use for Parkinson's disease, and their effect on symptoms
Demographics questionnaire | through study completion, an average of 2 weeks
  14-item questionnaire on demographic parameters
Diet questionnaire | through study completion, an average of 2 weeks
  18-item questionnaire on diet
Prevalence of increased COMT activity in urine | through study completion, an average of 2 weeks
  Catechol-O-methyltransferase

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc Centre of Expertise for Parkinson & Movement Disorders, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No